CLINICAL TRIAL: NCT06864442
Title: A Randomized Controlled Trial Comparing the Efficacy of Thread Embedding and Electroacupuncture in Speech-Language Rehabilitation in Patients With Post-Stroke Aphasia
Brief Title: Thread Embedding vs. Electroacupuncture for Post-Stroke Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loc Cong Dai Tran, MD (Other)
Collaborators: School of Medicine - Vietnam National University at Ho Chi Minh city (Other); Traditional Medicine Hospital at Dak Lak Province (Unknown)
Responsible Party: Sponsor-Investigator, Loc Cong Dai Tran, MD, Medical Doctor, Master of Sciences, School of Medicine - Vietnam National University at Ho Chi Minh city
Organization: School of Medicine - Vietnam National University at Ho Chi Minh city (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 793/HĐĐĐ-ĐHYD
Record Dates: First submitted 2025-03-02; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Post-stroke Aphasia
Keywords: Aphasia; Stroke; Catgut Thread Embedding; Electroacupuncture; Speech-Language Rehabilitation
MeSH Terms: conditions — Aphasia; Stroke | interventions — Electroacupuncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cagut Thread Embedding Group (Experimental): Patients received catgut thread embedding at day 0, day 10 and day 20.
  Interventions: Procedure: Catgut Thread Embedding
- Electroacupuncture Group (Active Comparator): Patients received daily electroacupuncture for 20 minutes over 30 days.
  Interventions: Procedure: Electroacupuncture

INTERVENTIONS:
Procedure: Catgut Thread Embedding — Catgut Thread Embedding involved implanting chromic catgut size 4.0 thread, which is attached to a 23G guide needle, into subcutaneous tissue at EX-HN21 acupoint. The guide needle was removed after insertion, while the thread remained and dissolved over 10-15 days to provide continuous stimulation.
  Other Names: Thread Embedding; Catgut Embedding
  Arms: Cagut Thread Embedding Group
Procedure: Electroacupuncture — Electroacupuncture was administered using four needles (0.3 × 25 mm, diameter × length) inserted at GV-20, EX-HN21, external EX-HN12, and external EX-HN13 acupoints. Electrical stimulation was delivered via the KWD-808I Multipurpose Health Device (Changzhou Yingdi Electronic Medical Device Co., China) with parameters set at 3 Hz frequency and 0.6 ms pulse width, the intensity was adjusted according to the patient's perception. Electroacupuncture was performed daily, except on Saturdays, Sundays, and Vietnamese national holidays, over a treatment course of 30 days.
  Other Names: Electrical Acupuncture; Electrical Stimulation Acupuncture
  Arms: Electroacupuncture Group

SUMMARY:
The goal of this clinical trial was to learn if thread embedding or electroacupuncture can treat language function impairment in patients with post-stroke aphasia, a condition affecting communication after a stroke. The main questions it aimed to answer were:

Does thread embedding improve overall language function more effectively than electroacupuncture, as measured by the Goodglass and Kaplan Aphasia Severity Rating Scale (ASRS)? How do thread embedding and electroacupuncture compare in improving specific language skills, such as motor speech, sensory language, reading, and naming, as assessed by the Boston Diagnostic Aphasia Examination (BDAE)? Researchers compared thread embedding (TE group) to electroacupuncture (EA group) to see if thread embedding provides better or similar effects on language recovery.

Participants:

Underwent a 30-day intervention with language assessments at the start and end of the period.

Were randomly assigned to either the thread embedding group, receiving treatment every 10 days, or the electroacupuncture group, receiving daily 20-minute sessions.

DETAILED DESCRIPTION:
This study was designed as a randomized, open-label, parallel-group trial conducted at the Traditional Medicine Hospital in Dak Lak, Vietnam. It received ethical approval from the Biomedical Research Ethic Committee at the University of Medicine and Pharmacy at Ho Chi Minh City (Approval No. 739/HĐĐĐ-ĐHYD, dated December 14, 2021). The interventions were delivered by certified traditional medicine practitioners following strict protocols (STRICTA 2010).

Catgut Thread Embedding (TE group): Participants received thread embedding at the EX-HN21 acupoint.

Electroacupuncture (EA group): Participants underwent daily 20-minute sessions in 30 days.

Language function was assessed using standardized tools, and data were analyzed with R. Statistical tests (chi-square, t-tests) compared baseline characteristics and outcomes, with a significance level of p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with post-stroke aphasia (severity levels 0-4 on the Goodglass and Kaplan scale)
* Aged 18 years or older
* Fluent in Vietnamese
* Alert and mentally competent (no psychiatric or neurological disorders affecting communication)
* No pre-existing speech or language disorders
* Willing to participate and provide signed informed consent
* Treated as inpatients at the Traditional Medicine Hospital, Dak Lak

Exclusion Criteria:

* Severe physical exhaustion or skin ulcers/infections at intervention sites
* Presence of a pacemaker
* Allergy to catgut threads
* Post-stroke patients awaiting cranioplasty
* Complex disease progression requiring alternative treatments during the study (data analyzed as treatment failures)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Boston Diagnostic Aphasia Examination (BDAE) | Day 0 and Day 30
  The Boston Diagnostic Aphasia Examination (BDAE) is a comprehensive and standardized tool designed to evaluate specific language functions in individuals with aphasia. It provides detailed insights into various language domains, including:
  Motor speech: Assesses articulation and fluency. Sensory language: Evaluates comprehension of spoken language. Reading skills: Measures the ability to read and understand written text. Naming skills: Tests the ability to name objects or concepts.
  Each domain is scored on a scale from 0 to 4, where:
  0: Indicates severe impairment (e.g., complete inability to speak or comprehend).
  4: Reflects mild or no impairment (near-normal language function). In practice, the BDAE is administered through structured tasks such as picture naming, sentence repetition, auditory comprehension tests, and reading exercises.
Goodglass and Kaplan's Aphasia Severity Rating Scale (ASRS) | Day 0 and Day 30
  The Goodglass and Kaplan's Aphasia Severity Rating Scale (ASRS) is a widely used tool that assesses the overall severity of aphasia. It employs a single scale ranging from 0 to 5 to summarize the general impact of aphasia on a patient's communication abilities:
  0: Very severe aphasia (e.g., no meaningful speech or comprehension). 1-2: Severe aphasia (e.g., limited speech and poor comprehension). 3-4: Moderate to mild aphasia (e.g., functional communication with noticeable deficits).
  5: Minimal or no aphasia (near-normal language function). The ASRS is typically scored based on clinical observation and interaction with the patient, focusing on their performance in everyday communication tasks like spontaneous speech, following commands, and answering questions.

SECONDARY OUTCOMES:
Adverse Events of Thread Embedding | Throughout the 30-day intervention period
  Incidence of adverse events (e.g., bleeding, infection, needle shock) monitored clinically during and after the intervention period.

OTHER OUTCOMES:
Baseline Characteristics | Day 0
  Baseline data were collected through patient interviews, medical records, and diagnostic tests. Demographic variables included age, categorized as ≤49, 50-69, or ≥70 years, gender, and education level, ranging from primary to post-secondary. Comorbid conditions were assessed as follows: hypertension was identified by blood pressure ≥140/90 mmHg or use of antihypertensive drugs, cardiovascular disease was determined by patient history and ECG results, diabetes was diagnosed if HbA1c ≥6.5%, fasting glucose ≥126 mg/dL, 2-hour glucose ≥200 mg/dL, random glucose ≥200 mg/dL with symptoms, or if patients were on diabetes medication, and dyslipidemia was confirmed by LDL ≥160 mg/dL, HDL <40 mg/dL, triglycerides ≥200 mg/dL, or total cholesterol ≥240 mg/dL. Stroke-related details encompassed the type, either hemorrhagic or ischemic, time since stroke, classified as ≤1 month or >1 month, and recurrence, noted as first-time or recurrent.

CONTACTS AND LOCATIONS:
Overall Officials: Minh-Anh Ngo Le Nguyen, Doctor of Philosophy, Study Chair — University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City, Vietnam; Linh Anh Truong, Master of Science, Study Director — Tay Nguyen University, Buon Ma Thuot City, Dak Lak Province, Vietnam
Locations (1):
- Traditional Medicine Hospital, Buon Ma Thuot, Dak Lak, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided
No specific plan is outlined in the document. A decision on sharing individual participant data (e.g., demographic characteristics, language assessment scores) will be determined when the article published, based on institutional policies and ethical considerations.
  Directly contact the corresponding author for more information.

REFERENCES:
- [Background] Sinanovic O, Mrkonjic Z, Zukic S, Vidovic M, Imamovic K. Post-stroke language disorders. Acta Clin Croat. 2011 Mar;50(1):79-94. PMID 22034787
- [Background] Mazaux JM, Lagadec T, de Seze MP, Zongo D, Asselineau J, Douce E, Trias J, Delair MF, Darrigrand B. Communication activity in stroke patients with aphasia. J Rehabil Med. 2013 Apr;45(4):341-6. doi: 10.2340/16501977-1122. PMID 23468019
- [Background] Gerstenecker A, Lazar RM. Language recovery following stroke. Clin Neuropsychol. 2019 Jul;33(5):928-947. doi: 10.1080/13854046.2018.1562093. Epub 2019 Jan 30. PMID 30698070
- [Background] Lazar RM, Speizer AE, Festa JR, Krakauer JW, Marshall RS. Variability in language recovery after first-time stroke. J Neurol Neurosurg Psychiatry. 2008 May;79(5):530-4. doi: 10.1136/jnnp.2007.122457. Epub 2007 Sep 10. PMID 17846113
- [Background] Berthier ML, Garcia-Casares N, Walsh SF, Nabrozidis A, Ruiz de Mier RJ, Green C, Davila G, Gutierrez A, Pulvermuller F. Recovery from post-stroke aphasia: lessons from brain imaging and implications for rehabilitation and biological treatments. Discov Med. 2011 Oct;12(65):275-89. PMID 22031666